CLINICAL TRIAL: NCT01716065
Title: Impact of Regional Anesthesia Versus General Anesthesia on Immune Modulation and Clearance of Circulating Tumor Cells (CTC) in Subjects Undergoing Surgery for Primary Nonmetastatic Breast Cancer
Brief Title: Regional Anesthesia Versus General Anesthesia on Circulating Tumor Cells (CTC)
Acronym: CTC
Status: Completed | Type: Observational
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Other Study IDs: 355841-17
Record Dates: First submitted 2012-10-17; First posted 2012-10-29 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer
Keywords: Anesthesia, Circulating tumor cells
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples collected for CTC analysis (2 tubes of 8ml of blood) will be drawn at 4 time points: pre-operative (at least 24 hours before surgery), immediate prior to surgery, 12-24 hours post-operative, and 5-7 days post-operative.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine whether the type of anesthesia during breast cancer surgery has any impact on the way a patient's immune system functions for a brief period after surgery. If the investigators find that one type of anesthesia versus the other is more beneficial to a patient's immune system, then the investigators may use this information to design a larger study to exam the effect of anesthesia better.

DETAILED DESCRIPTION:
There are two different types of anesthesia that the investigators can use for subjects undergoing breast surgery. The first type is called "general anesthesia" (GA) which is when a person "goes to sleep" with a breathing tube and then receives intravenous (IV) pain medicine during and after surgery to minimize surgical pain. The other type of anesthesia is called "regional anesthesia" (RA), or "nerve blocks" which numb up the nerves that supply the breast area. By doing this type of anesthesia, subjects often don't go "to sleep" with a breathing tube, instead, they get heavy IV sedation and take a "deep nap" during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects should be over 18 years of age and capable of providing informed consent indicating awareness of the investigational nature of this trial, in keeping with institutional policy
* Written informed consent must be obtained from each subject prior to entering the study
* Subjects with primary non-metastatic AJCC stages I, II or III, scheduled to undergo either unilateral mastectomy with or without Sentinel lymph node biopsy or axillary dissection, or unilateral lumpectomy with Sentinel lymph node biopsy or axillary lymph node dissection
* Able to stay overnight in the hospital post surgery

Exclusion Criteria:

* Any subject younger than 18 years or older than 85 years of age
* History of previous breast surgery (aside from biopsy), planned breast conserving operation (isolated lumpectomy) or reconstruction (rectus or latissimus flap)
* American Society of Anesthesia (ASA) classification of 4 or greater, or any contraindication to having regional anesthesia
* Any subjects who receives an intraoperative or postoperative blood transfusion during the period of venous blood sampling
* Subjects who are pregnant. Exclusion of the possibility of pregnancy by testing (urine HCG) or by history (tubal ligation, hysterectomy, or menopause) is required prior to inclusion in the study
* Subjects with active infectious process at the site of proposed paravertebral injection
* Subjects with significant allergy to local anesthetics
* Subjects who convert from RA to GA during surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll female and male military health care beneficiaries between the ages 18-85 years old presenting with the diagnosis of primary non-metastatic breast cancer, American Joint Committee on Cancer (AJCC) Stages I, II or III, undergoing surgery with curative intent
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Circulating Tumor Cells | 5 days
  blood will be drawn preoperative( at least 24 hours before surgery), immediate prior to surgery, immediately postoperative, 12-24 hours postoperative, and at postoperative appointment

SECONDARY OUTCOMES:
Levels of cytokines | 5 days
breast cancer antibodies | 5 days
Dendritic Cells | 5 days
T and B lymphocytes | 5 days
Natural Killer Cells (NK cells) | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States